CLINICAL TRIAL: NCT05631665
Title: Evaluation of Sexual Functions After Non-ablative Er:Yag Genital Laser Treatment in Postmenopausal Patients
Brief Title: Genital Laser Treatment in Postmenopausal Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Pınar Kadirogulları, Pinar KADIROGULLARI Assoc.Prof, Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATADEK/2022.11
Record Dates: First submitted 2022-11-04; First posted 2022-11-30 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Dyspareunia; Menopause; Sexual Activity; Atrophy Vulva
Keywords: Fractional CO2 Laser; Vaginal Dryness; Vulvovaginal Atrophy
MeSH Terms: conditions — Dyspareunia; Sexual Behavior

STUDY DESIGN:
Intervention Model Description: Patients who are in the postmenopausal period and undergo laser treatment for sexual problems
Masking Description: The group of patients who are in the postmenopausal period and undergo laser treatment for sexual problems.
  Laser will be applied to the postmenopausal patient group with vaginal dryness and dyspareunia complaints. This group will form the study group. The same surveys will be made before and after the procedure in the 1st month, 3rd month and 6th month. According to the results of the survey, the rate of improvement in sexual problems will be studied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- postmenopausal women (Experimental): women with postmenopausal sexual function problems will be the study arm
  Interventions: Other: Survey results before and after laser treatment

INTERVENTIONS:
Other: Survey results before and after laser treatment — Determination of sexual activity rates as points with a questionnaire before and after laser treatment for patients with postmenopausal sexual function problems.

SUMMARY:
Regulation of sexual functions without hormonal support in order to correct the sexual dysfunctions in women with the estrogen hormone lost in the menopausal process. Recently, the reaction to hormonal treatments and the fact that patients with a family history of breast cancer or gynecological cancer cannot receive hormonal treatment have been the reason for applying to alternative treatments. Lubricant treatments are among the treatments that patients have compliance problems in the long term and avoid due to the difficulty of application.

Correcting female sexual dysfunctions and post-menopausal women's right to want to feel sexually healthy are the most natural rights.

Because sexual dysfunctions cause physiological and psychological problems in women. Thanks to the laser treatment, it is aimed to eliminate the atrophy and sexual dysfunctions of women, thanks to the application of approximately 2 sessions without the need for long-term medication.

DETAILED DESCRIPTION:
The genitourinary syndrome of menopause (GSM) is a physiological process that affects more than 50% of postmenopausal women. It is a new definition that defines lower genital and urinary tract symptoms due to decreased estrogen levels in the menopausal transition and postmenopausal period. At the anatomical and histological level, estrogens can determine retraction of the introitus, thinning and regression of the labia, prominence of the urethral meatus, thinning of the vaginal epithelium and lamina propria layers with decreased glycogen stores, reduction in the papillae, and vascularization. Common symptoms of GSM include vaginal burning, itching, dryness, decreased lubrication, irritation, and dyspareunia. It may also include urinary symptoms such as urgency and dysuria.

Vaginal moisturizers, continuous sexual activity and lubricants are recommended as first-line treatment by the North American Menopause Society and The Endocrine Society in the treatment of GSM. When these first-line treatments are inadequate, local estrogen therapy or selective estrogen receptor modulators may be considered for suitable candidates. According to the International Urogynecological Association document, low-dose vaginal estrogens resulted in a level of evidence 1 for safe and effective treatment of GSM symptoms. In the last few years, increasing research has focused on alternative treatments such as energy-based devices and the use of laser (i.e., fractional microablative CO2, Er:YAG laser) while various studies are reassuring about the side effects of these treatments, long-term side effects remain to be defined. Previous studies have shown that fractional carbon dioxide (CO2) laser is effective and safe in improving vaginal symptoms associated with GSM. The use of this device should be done safely by trained health professionals, with certified devices, in exact indications, ideal conditions according to contraindications. The aim of the study was to evaluate the efficacy of laser therapy with CO2 vaginal laser on GSM symptoms with a prospective approach based on quality of life questionnaires completed by treated patients.

ELIGIBILITY:
Inclusion Criteria:

* female patients in menopause
* have not received previous treatment for sexual problems
* not receiving hormone therapy
* cancer vs. with no history of chemotherapy or radiotherapy
* patients with sound cognitive functions who can answer the questionnaire questions

Exclusion Criteria:

* menstruating
* cancer treatment recipients
* hormone users --those who do not have sexual activity

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
survey results before laser treatment | 6 months
  Determination of sexual activity rates as points by questionnaire before laser procedure in patients with postmenopausal sexual function problems : Scoring will be done based on survey responses.
  Sexual Function Index (FSFI) scoring will be used.The FSFI questionnaire consists of 19 questions; It evaluates 6 main factors as sexual desire, sexual arousal, lubrication, orgasm, satisfaction and pain/discomfort. The highest total raw score that can be obtained in this scale is 95, the lowest raw score is 4, and the highest score is 36 and the lowest score is 2 after multiplying the coefficients.
survey results after laser treatment | 6 months
  Determination of sexual activity rates as points by questionnaire after laser procedure in patients with postmenopausal sexual function problems.Scoring will be done based on survey responses.
  Sexual Function Index (FSFI) scoring will be used.The FSFI questionnaire consists of 19 questions; It evaluates 6 main factors as sexual desire, sexual arousal, lubrication, orgasm, satisfaction and pain/discomfort. The highest total raw score that can be obtained in this scale is 95, the lowest raw score is 4, and the highest score is 36 and the lowest score is 2 after multiplying the coefficients.

CONTACTS AND LOCATIONS:
Locations (1):
- Acıbadem University Atakent Hospital, Department of Obstetrics and Gynecology,, Istanbul, Turkey (Türkiye)